CLINICAL TRIAL: NCT03875053
Title: Evaluation of Obstructive Sleep Apnea in Head and Neck Cancer
Brief Title: Home Sleep Apnea Machine in Evaluating Obstructive Sleep Apnea in Patients With Stage III-IV Head and Neck Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No accrual
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Ammar Sukari, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-135; P30CA022453 (NIH)
Record Dates: First submitted 2019-02-11; First posted 2019-03-14 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-10

CONDITIONS: Locally Advanced Head and Neck Squamous Cell Carcinoma; Metastatic Head and Neck Squamous Cell Carcinoma
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Monitoring, Physiologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Monitoring device, Quality of Life Assessment, Questionnaire (Experimental): Patients wear the home sleep apnea machine overnight. Patients undergoing standard of care CRT wear the home sleep apnea machine a second time 3 months after completion of CRT.
  Interventions: Diagnostic Test: Monitoring Device; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Diagnostic Test: Monitoring Device — Patients wear the home sleep apnea machine overnight. Patients undergoing standard of care CRT wear the home sleep apnea machine a second time 3 months after completion of CRT.
  Other Names: Monitor
Other: Quality-of-Life Assessment — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This trial studies information from a home sleep apnea machine to evaluate obstructive sleep apnea in patients with stage III-IV head and neck cancer. Sleep apnea (trouble breathing during sleep) can occur in head and neck cancer patients who have swelling in their neck. Wearing a sleep apnea machine overnight may help doctors evaluate obstructive sleep apnea in patients with head and neck cancer.

DETAILED DESCRIPTION:
This is a single center study in HNSCC subjects to assess the effects of CRT on OSA.. Patients will be screened with a physical exam and questionnaire (The Berlin questionnaire, STOP-BANG, PSQI) and when eligible, will have the home sleep study (Specific aim 1). The low risk group (based on the physical exam and questionnaire) with stage IVc will not be eligible for the home sleep study and will concentrate on palliation of their symptoms. For locally advanced HNSCC patients undergoing definitive CRT, post CRT home sleep study results will also be assessed (Specific aim 2). When the patient is diagnosed with OSA based on the home sleep study, or if the home sleep study is negative but if the patient had high risks based on the screening process, the patient will be referred to the sleep medicine clinic. If life-threatening obstructive sleep apnea is found, the patient will be referred to sleep medicine clinic right away and will be taken off study. Otherwise, the patients will prioritize their definitive CRT for HNSCC, and will be referred to sleep medicine clinic once CRT has been completed.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced (stage III-IVb) and metastatic (stage IVc) HNSCC who are referred to medical oncology. Patients may not have received upfront definitive surgical resection of the primary tumor or upfront neck dissection.
* Patients must be able to operate the home sleep study device.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2.

Exclusion Criteria:

* Patients should not have received any prior systemic chemotherapy or radiation therapy for locally advanced or metastatic HNSCC.
* Patients with tracheostomy or those requiring the assistance of a ventilator will be ineligible for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-25 (Estimated); Primary Completion 2023-08-24 (Estimated); Study Completion 2024-08-24 (Estimated)

PRIMARY OUTCOMES:
Obstructive sleep apnea (OSA) rate before and after chemoradiation therapy (CRT) in stage III-IVb patients undergoing CRT | Up to 1 year
  The definition of OSA will be defined as apnea-hypopnea index of > 5 for both pre and post CRT. The OSA rate is the proportion of patients diagnosed with OSA. Will be assessed using a two-sided McNemar test based on the OSA occurrence (Yes versus [vs.] No) for each patient. The OSA rates pre and post CRT will be described by means and their two-sided confidence intervals (Cls). The univariable and multivariable conditional logistic regression models will be further used for the primary objective with patients' baseline characteristics as covariates.

SECONDARY OUTCOMES:
Response to CRT | Up to 1 year
  Will be evaluated using Response Evaluation Criteria in Solid Tumors version 1.1. Will be described by mean and the two-sided CI. The univariable and multivariable binary (multinomial) logistic regression models will be used to assess the association of the effects of patients' baseline characteristics and the occurrence of OSA on the CRT responses.
Occurrence of OSA in stage III-IVb patients undergoing CRT | Up to 1 year
  Will be grouped into four categories (Yes/Yes, Yes/No, No/Yes, and No/No for pre/post CRT). Then a 2x4 contingency table will be generated by CRT response (binary; Yes vs. No) and OSA occurrence (quaternary; Yes/Yes vs. Yes/No vs. No/Yes vs. No/No) and a Chi- 23 squared test (or Fisher's exact test) will be used. The univariable and multivariable binary (multinomial) logistic regression models will be used to assess the association of the effects of patients' baseline characteristics and the occurrence of OSA on the CRT responses.
OSA rate in locally advanced or metastatic stage head and neck squamous cell carcinoma (HNSCC) patients | Up to 1 year
  A descriptive analysis will be performed on all patients enrolled and on all eligible patients who undergo home sleep apnea study to evaluate the OSA rate in locally advanced or metastatic stage HNSCC patients. The OSA rate will be estimated for locally advanced or metastatic stage HNSCC patients who enter the study in Part 1 and then will be described by mean and the two-sided Cl.

OTHER OUTCOMES:
Adherence rate to OSA treatment to 30 days | Up to 1 year
  It is defined as the ratio of the number of days adhered to OSA treatment to 30 days.
Incidence rate of OSA by MRI neck findings | Up to 1 year
  It is the OSA rate detected by MRI neck findings among oropharyngeal cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ammar Sukari, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (1):
- Barbara Ann Karmanos Cancer Institute, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No